CLINICAL TRIAL: NCT07124962
Title: Comparison of Post Operative Pain and Periapical Healing Following Regenerative Endodontics Using Platelet Rich Plasma vs Conventional Root Canal Treatment in Mature Single Rooted Teeth
Brief Title: PRP Regenerative Endodontics vs. Root Canal Treatment for Post-Op Pain and Healing in Mature Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HITEC-Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, fatimaharshad, Principal investigator, HITEC-Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dr Fatimah Arshad
Record Dates: First submitted 2025-08-11; First posted 2025-08-15 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Irreversible Pulpitis With Apical Periodontitis
MeSH Terms: interventions — Root Canal Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two treatment groups in parallel. Each participant will receive either regenerative endodontic treatment using platelet-rich plasma (PRP) or conventional root canal treatment (RCT). Both groups will be treated and followed simultaneously, and outcomes including post-operative pain and periapical healing will be compared between groups. No crossover or switching of interventions will occur.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Root Canal Treatment (RCT) (Active Comparator): Patients will undergo conventional root canal therapy, including canal preparation using hand k-files (#10-#45), irrigation with 3% sodium hypochlorite, and obturation using lateral condensation technique with resin-based sealer. The access cavity will be restored using Glass Ionomer Cement.
  Interventions: Procedure: Root Canal Therapy
- PRP Revascularization (Experimental): After canal disinfection and removal of double antibiotic paste, PRP derived from autologous blood will be injected into the canal space after inducing bleeding through over-instrumentation. A layer of Mineral Trioxide Aggregate (MTA) will be placed, followed by temporary GIC and final composite restoration after 7 days.
  Interventions: Procedure: Platelet-Rich Plasma (PRP) Revascularization

INTERVENTIONS:
Procedure: Root Canal Therapy — Regenerative endodontic procedure using autologous platelet-rich plasma injected into the root canal space to promote pulp-dentin regeneration, followed by placement of MTA and composite restoration.
  Arms: Conventional Root Canal Treatment (RCT)
Procedure: Platelet-Rich Plasma (PRP) Revascularization — Regenerative endodontic procedure using autologous platelet-rich plasma injected into the root canal space to promote pulp-dentin regeneration, followed by placement of MTA and composite restoration.
  Arms: PRP Revascularization

SUMMARY:
This randomized clinical trial aims to compare the effectiveness of regenerative endodontic treatment using platelet-rich plasma (PRP) with conventional root canal treatment (RCT) in mature single-rooted teeth diagnosed with irreversible pulpitis and periapical lesions. The primary outcomes assessed will be post-operative pain and periapical healing. A total of 46 patients will be randomly assigned to either the PRP group or the RCT group. Pain will be recorded at baseline, 24, and 48 hours post-operatively using a numerical rating scale. Periapical healing will be evaluated clinically and radiographically at 1 and 6 months using the Periapical Index (PAI). The study aims to determine whether PRP-based regenerative therapy offers superior outcomes compared to conventional root canal therapy.

DETAILED DESCRIPTION:
This randomized clinical trial is designed to evaluate and compare the clinical efficacy of regenerative endodontics using platelet-rich plasma (PRP) versus conventional root canal treatment (RCT) in mature single-rooted permanent teeth diagnosed with irreversible pulpitis and radiographic signs of periapical pathology (PAI score 4).

Recent advancements in regenerative endodontics have demonstrated the potential for biologically-based procedures that not only disinfect the root canal system but also aim to regenerate the pulp-dentine complex and promote periapical healing. Platelet-rich plasma (PRP), a natural autologous scaffold derived from the patient's blood, contains growth factors such as PDGF, IGF, TGF-β, and EGF that enhance tissue healing, angiogenesis, and stem cell proliferation.

This trial will enroll 46 patients aged 16-50 years, who will be randomly allocated into two groups:

Group A (Control Group): Will undergo standard two-visit conventional RCT using lateral condensation technique and resin-based sealer.

Group B (Intervention Group): Will receive regenerative endodontic therapy using PRP revascularization. After canal disinfection with double antibiotic paste, bleeding will be induced, and PRP will be placed in the canal, followed by MTA and restoration.

Pain intensity will be assessed using the Numerical Rating Scale (NRS) at baseline, 24, and 48 hours postoperatively. Periapical healing will be evaluated clinically and radiographically at 1 month and 6 months using the Periapical Index (PAI). Treatment success will be defined as the absence of clinical symptoms and radiographic evidence of healing or reduction in PAI score.

The study aims to determine whether PRP-based regenerative endodontics can reduce post-operative pain more effectively and promote faster and better periapical healing compared to conventional root canal therapy in mature teeth.

ELIGIBILITY:
Inclusion Criteria:

* Mature single rooted teeth diagnosed with irreversible pulpitis presenting with radiographic signs of periapical lesions (PAI score 4)
* Patients that fall in the ages between 16-50 years

Exclusion Criteria:

* Pregnant females
* Patients reporting with bruxism
* Teeth with severely curved canals
* Teeth with developmental anomalies, pathologic mobility, root fracture or a probing depth of >3mm
* Any allergy to medications or antibiotics (necessary to complete the procedure)

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Post-operative Pain Score | 24 hours and 48 hours after second treatment visit
  Patients will self-report pain levels on a 0-10 numerical rating scale, categorized as:
  0 = no pain 1-3 = mild pain 4-6 = moderate pain 7-10 = severe pain Pain will be assessed by phone call at 24 and 48 hours after the second visit.

SECONDARY OUTCOMES:
Periapical Healing Based on Periapical in Score | 1 month and 6 months post-treatment
  Healing is evaluated using the Periapical Index (PAI) based on radiographs taken with the Digora system. Improvement in PAI score from baseline indicates periapical healing. Treatment is considered successful if the tooth is asymptomatic, not tender to percussion, shows no swelling, and demonstrates radiographic healing.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Beenish Qureshi, BDS, FCPS, Study Chair — HITEC-Institute of Medical Sciences
Locations (1):
- Dental hospial, Hitec-IMS, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahmed YE, Ahmed GM, Ghoneim AG. Evaluation of postoperative pain and healing following regenerative endodontics using platelet-rich plasma versus conventional endodontic treatment in necrotic mature mandibular molars with chronic periapical periodontitis. A randomized clinical trial. Int Endod J. 2023 Apr;56(4):404-418. doi: 10.1111/iej.13886. Epub 2023 Jan 12. PMID 36565044